CLINICAL TRIAL: NCT01155635
Title: Carvedilol Post-intervention Long-term Administration in Large-scale Randomized Controlled Trial
Brief Title: Carvedilol Post-intervention Long-term Administration in Large-scale Trial
Acronym: CAPITAL-RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-417
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Adrenergic beta-Antagonists; Percutaneous coronary intervention
MeSH Terms: conditions — Myocardial Infarction | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beta-blocker (Active Comparator): Use of Carvedilol with any dose
  Interventions: Drug: Carvedilol
- Non Beta-blocker (Active Comparator): No use of Carvedilol
  Interventions: Drug: No Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Use of Carvedilol with any dose
  Arms: Beta-blocker
Drug: No Carvedilol — No use of Carvedilol
  Arms: Non Beta-blocker

SUMMARY:
The purpose of this study is to evaluate whether beta-blocker therapy improves 6-year clinical outcomes in patients with ST-segment elevation acute myocardial infarction and preserved left ventricular ejection fraction after primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Beta-blocker therapy is recommended after ST-segment elevation acute myocardial infarction (STEMI) in the current guidelines although its efficacy in those patients who have undergone primary percutaneous coronary intervention (PCI) has not been adequately evaluated. The purpose of this study is to evaluate whether beta-blocker, carvedilol improves 6-year clinical outcomes in patients with STEMI and preserved left ventricular ejection fraction after primary PCI. The design of this study is multicenter, open-label, randomized controlled trial enrolling 1300 patients without any exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI after primary PCI
* Patients with left ventricular ejection fraction more than or equal to 40%

Exclusion Criteria:

* Patients with left ventricular ejection fraction less than 40%
* Patients with contraindication for beta-blocker
* Patients with implantable cardioverter defibrillators
* Patients with end-stage malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2010-07; Primary Completion 2015-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 6-year
  Death from any reason
Composite of death, myocardial infarction, acute coronary syndrome, heart failure hospitalization | 6-year

SECONDARY OUTCOMES:
Cardiac death | 6-year
Sudden cardiac death | 6-year
Cardiovascular death | 6-year
Myocardial infarction | 6-year
Acute coronary syndrome | 6-year
Sustained ventricular tachycardia or ventricular fibrillation | 6-year
Heart failure hospitalization | 6-year
Stent thrombosis | 6-year
  Stent thrombosis defined by Academic Research Consortium
Target-vessel revascularization | 6-year
Clinically-driven target-lesion revascularization | 6-year
Any coronary revascularization | 6-year
Any clinically-driven coronary revascularization | 6-year
Coronary artery bypass grafting | 6-year
Stroke | 6-year
  Any ischemic and hemorrhagic strokes excluding transient ischemic attacks
Worsening of angina due to coronary spasm | 6-year
Bleeding complications | 6-year
  Bleeding complications defined by GUSTO and TIMI definitions
Composite of death, myocardial infarction, stroke, acute coronary syndrome, heart failure hospitalization, any coronary revascularization | 6-year
Composite of cardiac death, myocardial infarction, acute coronary syndrome, heart failure hospitalization | 6-year
Composite of cardiovascular death, myocardial infarction, stroke | 6-year

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Division of Cardiology, Kyoto University Hospital, Kyoto, Japan

REFERENCES:
- [Derived] Amano M, Izumi C, Watanabe H, Ozasa N, Morimoto T, Bingyuan B, Suwa S, Miyake M, Tamura T, Nakagawa Y, Kadota K, Inuzuka Y, Minamimoto Y, Furukawa Y, Kaji S, Suzuki T, Akao M, Inada T, Kimura T; CAPITAL-RCT Investigators. Effects of Long-Term Carvedilol Therapy in Patients With ST-Segment Elevation Myocardial Infarction and Mildly Reduced Left Ventricular Ejection Fraction. Am J Cardiol. 2023 Jul 15;199:50-58. doi: 10.1016/j.amjcard.2023.04.042. Epub 2023 May 26. PMID 37245250
- [Derived] Watanabe H, Ozasa N, Morimoto T, Shiomi H, Bingyuan B, Suwa S, Nakagawa Y, Izumi C, Kadota K, Ikeguchi S, Hibi K, Furukawa Y, Kaji S, Suzuki T, Akao M, Inada T, Hayashi Y, Nanasato M, Okutsu M, Kametani R, Sone T, Sugimura Y, Kawai K, Abe M, Kaneko H, Nakamura S, Kimura T; CAPITAL-RCT investigators. Long-term use of carvedilol in patients with ST-segment elevation myocardial infarction treated with primary percutaneous coronary intervention. PLoS One. 2018 Aug 28;13(8):e0199347. doi: 10.1371/journal.pone.0199347. eCollection 2018. PMID 30153268